CLINICAL TRIAL: NCT01161745
Title: PD-1/PD-L1 Pathway in T Lymphocyte Apoptosis and Monocyte Dysfunction in Septic Patients
Brief Title: PD-1/PD-L1 Pathway Study on Septic Patients
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Xiao-ming Deng, Department of Anesthesiology and Intensive Care Unit
Other Study IDs: ANETHDEPT-001
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-06

CONDITIONS: Sepsis
Keywords: sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — peripheral venous blood from septic patients and healthy controls, anticoagulate with EDTA-K2
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to identify that whether PD-1/PD-L1 pathway will change in human sepsis, and whether PD-1/PD-L1 pathway play an important role in sepsis induced immunosuppression.

DETAILED DESCRIPTION:
First, we will detect PD-L1 expression on PBMC of septic patients and healthy controls.

Second, blockade of PD-1/PD-L1 pathway in vitro and stimulate with some biomolecules and then analyze the PBMC function and apoptosis by flow cytometry.

Then, compare with healthy controls and find the differences.

ELIGIBILITY:
Inclusion Criteria:

* patients who develop sepsis

Exclusion Criteria:

* patients with cirrhosis or renal dysfunction
* patients with dyscrasia
* patients with autoimmunity diseases
* patients with severe cardiac and pulmonary diseases
* patients with hematological diseases
* patients with diabetes mellitus
* patients with malignant tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who develop sepsis
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-ming Deng, doctor, Principal Investigator — Changhai Hospital, the Second Military Medical University